CLINICAL TRIAL: NCT01315015
Title: Breast Cancer Screening With MRI in Women Aged 50-75 Years With Extremely Dense Breast Tissue: the DENSE Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Breast Cancer Screening Organisations (Unknown); Dutch Reference Centre for Screening (Unknown); National Institute for Public Health and the Environment (RIVM) (Other Government); The Netherlands Cancer Institute (Other); University Medical Center Nijmegen (Other); Jeroen Bosch Ziekenhuis (Other); Albert Schweitzer Hospital (Other); Hospital Group Twente (ZGT) (Unknown); Amsterdam UMC, location VUmc (Other); Maastricht University Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Dutch Cancer Society (Other); Pink Ribbon Inc. (Industry); A Sister's Hope (Other); Bayer (Industry); Stichting Kankerpreventie Midden-West (Unknown); Volpara Solutions (Other)
Responsible Party: Principal Investigator, C.H. van Gils, Professor of Clinical Epidemiology of Cancer, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UMCU DENSE; ZONMW-200320002-UMCU (Other Grant/Funding Number: ZonMw); Pink Ribbon-10074 (Other Grant/Funding Number: Dutch Pink Ribbon / a Sister's hope); BSP-DENSE (Other Grant/Funding Number: Bayer HealthCare, Medical Care); DCS-UU-2009-4348 (Other Grant/Funding Number: Dutch Cancer Society); DCS-UU-2014-6859 (Other Grant/Funding Number: Dutch Cancer Society); UMCU DENSE (Other Grant/Funding Number: University Medical Center Utrecht)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Breast neoplasm; Magnetic Resonance Imaging; Breast density; Early detection of cancer; Cancer screening test; Secondary prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Contrast enhanced breast MRI (Experimental): The additional MRI will take place biennially after the regular screening mammogram for a study period of 6 years.
  Interventions: Other: Contrast enhanced breast MRI
- Regular breast cancer screening (No Intervention): No further follow-up until next scheduled screening examination two years later (according to the current Dutch guideline).

INTERVENTIONS:
Other: Contrast enhanced breast MRI — Gadolinium contrast is administered as a bolus with a standard dose of 0.1 mL/kg followed by a saline flush of 30 mL.
  Other Names: MR Mammography
  Arms: Contrast enhanced breast MRI

SUMMARY:
The purpose of this study is to determine the cost-effectiveness of biennial screening with mammography and MRI compared to mammography alone in women aged 50-75 years and who show > 75% mammographic density.

DETAILED DESCRIPTION:
Women with very high mammographic density have a four to six fold higher breast cancer risk than women with low mammographic density. At the same time, the sensitivity of mammography is seriously impaired in women with high mammographic density, leading to many missed cases. Nevertheless, in the Netherlands this high risk group is currently screened between the age of 50 and 75 years with mammography only. MRI is likely to lead to better detection of breast tumors in women with high mammographic density, because it has a much higher sensitivity than mammography. The DENSE trial investigates the additional value of MRI for breast cancer screening in this risk group. Participants with extremely dense breasts (ACR4) and a negative mammogram are randomized to 'additional MRI' (n=7,237) versus 'current practice' (n=28,948).

ELIGIBILITY:
Inclusion Criteria:

* Dutch breast cancer screening participants, aged 50-75 years
* > 75% mammographic density
* Negative mammographic examination (BIRADS 1 or 2)

Exclusion Criteria:

Contraindications for MRI

* The presence of intracorporeal metals
* Adverse reaction to a (gadolinium-based) contrast agent in the past
* Severely impaired renal function (GFR < 40 mL/min)
* Pregnant or lactating women
* Claustrophobia
* Adiposity (> 150 kg)

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40373 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2023-04 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
The number of interval cancers will be compared between the MRI group and the control group | 8 years (with an interim analysis every two years; time period between two screening rounds)
  The intervention will be carried out for six years, i.e. 3 screening rounds. Given a two year recruitment period, the total study time will be 8 years.

SECONDARY OUTCOMES:
The number of MRI screen-detected tumors will be determined | 6 years (with an interim analysis every two years; time period between two screening rounds)
  The MRI examination will take place every two years (0, 2 and 4 years after inclusion). Given a two year recruitment period, the total study time will be 6 years.
Tumor size, stage and grade distributions, including their histological and molecular subtypes, diagnosed in both study groups will be compared | 8 years (with an interim analysis every two years; time period between two screening rounds)
  The intervention will be carried out for six years, i.e. 3 screening rounds. Given a two year recruitment period, the total study time will be 8 years.
The referral rate in the MRI study group will be determined | 6 years (with an interim analysis every two years; time period between two screening rounds)
  The MRI examination will take place every two years (0, 2 and 4 years after inclusion). Given a two year recruitment period, the total study time will be 6 years.
The positive predictive value (and the amount of false-positive diagnoses) of MRI will be determined using the histological diagnosis as the reference test | 6 years (with an interim analysis every two years; time period between two screening rounds)
  The MRI examination will take place every two years (0, 2 and 4 years after inclusion). Given a two year recruitment period, the total study time will be 6 years.
The number of biopsies per positive MRI will be determined | 6 years (with an interim analysis every two years; time period between two screening rounds)
  The MRI examination will take place every two years (0, 2 and 4 years after inclusion). Given a two year recruitment period, the total study time will be 6 years.
The mortality rate in the MRI group will be compared with the control group using the MISCAN computer simulation program | 8 years
  The intervention will be carried out for six years, i.e. 3 screening rounds. Given a two year recruitment period, the total study time will be 8 years.
The cost-effectiveness of MRI will be estimated using the MISCAN computer simulation program | 8 years
  The intervention will be carried out for six years, i.e. 3 screening rounds. Given a two year recruitment period, the total study time will be 8 years.
The impact of MRI screening on quality of life will be assessed using standardized and validated questionnaires | 8 years
  The intervention will be carried out for six years, i.e. 3 screening rounds. Given a two year recruitment period, the total study time will be 8 years.

CONTACTS AND LOCATIONS:
Overall Officials: Carla H van Gils, PhD, Principal Investigator — UMC Utrecht; Wouter B Veldhuis, MD PhD, Principal Investigator — UMC Utrecht
Locations (9):
- Netherlands (9):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Hospital Group Twente (ZGT), Almelo
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - VU University Medical Center, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Hospital Group Twente (ZGT), Hengelo
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] van Grinsven SEL, Mann RM, Monninkhof EM, Duvivier K, de Jong MDF, de Koekkoek-Doll PK, Loo CE, Pijnappel RM, van der Sluijs R, Veltman J, van Gils CH, Veldhuis WB; DENSE Trial Study Group. Multireader Diagnostic Accuracy of Abbreviated Breast MRI for Screening Women with Extremely Dense Breasts. Radiology. 2025 May;315(2):e241233. doi: 10.1148/radiol.241233. PMID 40392091
- [Derived] Verburg E, van Gils CH, van der Velden BHM, Bakker MF, Pijnappel RM, Veldhuis WB, Gilhuijs KGA. Validation of Combined Deep Learning Triaging and Computer-Aided Diagnosis in 2901 Breast MRI Examinations From the Second Screening Round of the Dense Tissue and Early Breast Neoplasm Screening Trial. Invest Radiol. 2023 Apr 1;58(4):293-298. doi: 10.1097/RLI.0000000000000934. Epub 2022 Oct 17. PMID 36256783
- [Derived] Verburg E, van Gils CH, van der Velden BHM, Bakker MF, Pijnappel RM, Veldhuis WB, Gilhuijs KGA. Deep Learning for Automated Triaging of 4581 Breast MRI Examinations from the DENSE Trial. Radiology. 2022 Jan;302(1):29-36. doi: 10.1148/radiol.2021203960. Epub 2021 Oct 5. PMID 34609196
- [Derived] Veenhuizen SGA, de Lange SV, Bakker MF, Pijnappel RM, Mann RM, Monninkhof EM, Emaus MJ, de Koekkoek-Doll PK, Bisschops RHC, Lobbes MBI, de Jong MDF, Duvivier KM, Veltman J, Karssemeijer N, de Koning HJ, van Diest PJ, Mali WPTM, van den Bosch MAAJ, van Gils CH, Veldhuis WB; DENSE Trial Study Group. Supplemental Breast MRI for Women with Extremely Dense Breasts: Results of the Second Screening Round of the DENSE Trial. Radiology. 2021 May;299(2):278-286. doi: 10.1148/radiol.2021203633. Epub 2021 Mar 16. PMID 33724062
- [Derived] Bakker MF, de Lange SV, Pijnappel RM, Mann RM, Peeters PHM, Monninkhof EM, Emaus MJ, Loo CE, Bisschops RHC, Lobbes MBI, de Jong MDF, Duvivier KM, Veltman J, Karssemeijer N, de Koning HJ, van Diest PJ, Mali WPTM, van den Bosch MAAJ, Veldhuis WB, van Gils CH; DENSE Trial Study Group. Supplemental MRI Screening for Women with Extremely Dense Breast Tissue. N Engl J Med. 2019 Nov 28;381(22):2091-2102. doi: 10.1056/NEJMoa1903986. PMID 31774954
- [Derived] de Lange SV, Bakker MF, Monninkhof EM, Peeters PHM, de Koekkoek-Doll PK, Mann RM, Rutten MJCM, Bisschops RHC, Veltman J, Duvivier KM, Lobbes MBI, de Koning HJ, Karssemeijer N, Pijnappel RM, Veldhuis WB, van Gils CH. Reasons for (non)participation in supplemental population-based MRI breast screening for women with extremely dense breasts. Clin Radiol. 2018 Aug;73(8):759.e1-759.e9. doi: 10.1016/j.crad.2018.04.002. Epub 2018 Jun 18. PMID 29759590

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study protocol (2011-06-07): https://cdn.clinicaltrials.gov/large-docs/15/NCT01315015/Prot_SAP_000.pdf